CLINICAL TRIAL: NCT05480319
Title: Prospective Deployment of a Cardiac Arrest Response System (EDICARS) in the Emergency Department: A Cluster Randomized Controlled Trial
Brief Title: Prospective Deployment of a Cardiac Arrest Response System (EDICARS) in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 202205061RINC
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDICARS (Experimental)
  Interventions: Other: EDICARS
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: EDICARS — The investigators propose to (1) Embed the EDICAS into our hospital information system (HIS) in real-time at ED triage to identify high-risk patients (EDICAS 6+); and (2) Distribute wearable smart wristbands to high-risk patients to augment vital signs monitoring and send alerts based on GBTM results. The detection and intervention components together form the rapid response system, the Emergency Department In-hospital Cardiac Arrest Response System (EDICARS).
  Arms: EDICARS
Other: Usual care — Usual care will be assigned to this arm. No additional interventions.
  Arms: Usual care

SUMMARY:
Based on data from the American Heart Association's (AHA) Get With the Guidelines-Resuscitation (GTWG-R) registry, the incidence of adult treated in-hospital cardiac arrest (IHCA) was about 10 per 1,000 bed-days (290,000 patients per year), and 15 to 20% of adult IHCA patients survived to hospital discharge (i.e., ~80% mortality). Despite the significant morbidity and mortality caused by IHCA, ED-based IHCA is surprisingly less studied. The investigators have utilized electronic medical record (EMR)'s big data (>700,000 visits) from our hospital to investigate, for the first time, the epidemiology and outcome of IHCA in the ED in Taiwan. The investigators also have developed and validated a simple prediction tool for ED-based IHCA, the Emergency Department In-hospital Cardiac Arrest Score (EDICAS). This tool has also been externally validated using Far Eastern Memorial Hospital's ED data. In addition, the investigators also have developed and validated a vital-sign trajectory-based longitudinal model (group-based trajectory modeling [GBTM]) to predict ED-based IHCA.

Based on these studies, the investigators now propose to (1) Embed the EDICAS into our hospital information system (HIS) in real-time at ED triage to identify high-risk patients (EDICAS 6+); and (2) Distribute wearable smart wristbands to high-risk patients to augment vital signs monitoring and send alerts based on GBTM results. The detection and intervention components together form the rapid response system, the Emergency Department In-hospital Cardiac Arrest Response System (EDICARS). In this study, the investigators will enroll and randomize 10 attending physicians into the EDICARS or the usual care arm for 3 months, with each of them treating 100 patients (patients clustered within physicians). The trial will stop for 2 months as a wash-out period, and an interim analysis will be performed. The physicians will then cross over, and each of them will treat 100 patients for another 3 months. A total of 2,000 adult patients will be enrolled. The primary outcome is a composite rate of ED-based IHCA and intensive care unit (ICU) admission. The secondary outcomes include time from ED triage to ED-based cardiac arrest, ICU and hospital length of stay, early ward-based IHCA, and early ICU transfer.

ELIGIBILITY:
Inclusion Criteria:

* ED patients aged 20 years at recruitment

Exclusion Criteria:

* Inability to sign informed consent;
* Diagnosis of psychiatric disorders that would limit the ability to comply with the study protocol (e.g., wearing a wristband);
* Intending to leave ED against medical advice;
* Already enrolled or planning to enroll in a research study that would conflict with full participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2010 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
ED-based in-hospital cardiac arrest (IHCA) and intensive care unit (ICU) admission. | During the stay in the emergency department, a median length of 3 hours
  The primary outcome is a composite rate of ED-based IHCA and intensive care unit (ICU) admission.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan